CLINICAL TRIAL: NCT03552835
Title: Management of Occlusal Dentinal Caries in Deciduous Molars- A Clinical and Radiographic Evaluation of Three Approaches
Brief Title: Management of Occlusal Dentinal Caries in Deciduous Molars
Acronym: MOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sneha D. Suwarnkar (Other)
Responsible Party: Sponsor-Investigator, Sneha D. Suwarnkar, Principal investigator, Saraswati-Dhanwantari Dental College & Hospital
Organization: Saraswati-Dhanwantari Dental College & Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SarswatiDhanwantari
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Caries, Dental
Keywords: no caries removal; partial caries removal upto soft dentin; partial caries removal upto firm dentin
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: occlusal dentinal caries were managed by either partial caries removal upto soft dentin or partial caries removal upto firm dentin or no caries removal and were compared
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no caries removal (Experimental): mandibular occlusal caries were treated with placement of stainless steel crown with no caries removal
  Interventions: Procedure: no caries removal
- partial caries removal upto soft dentin (Experimental): mandibular occlusal caries were treated by partial caries removal upto soft dentin
  Interventions: Procedure: partial caries removal upto soft dentin
- partial caries removal upto firm dentin (Experimental): mandibular occlusal caries were treated by partial caries removal upto firm dentin
  Interventions: Procedure: partial caries removal upto firm dentin

INTERVENTIONS:
Procedure: no caries removal — occlusal caries were treated with no caries removal and placement of stainless steel crown
  Arms: no caries removal
Procedure: partial caries removal upto soft dentin — occlusal caries were treated by partial caries removal upto soft dentin followed by Glass Ionomer Cement placement as a base and composite restoration
  Arms: partial caries removal upto soft dentin
Procedure: partial caries removal upto firm dentin — occlusal caries were treated by partial caries removal upto firm dentin followed by Glass Ionomer Cement placement as a base and composite restoration
  Arms: partial caries removal upto firm dentin

SUMMARY:
This study evaluated and compared the efficacy of no caries removal and sealing with a well-adapted and crimped stainless steel crown verses selective caries removal upto soft dentin and upto firm dentin in healing and/or preventing progression of moderate to deep occlusal dentinal caries.

DETAILED DESCRIPTION:
Dental caries is a complex multifactorial disease and is one of the most prevalent diseases throughout history. It can cost a lot of money to treat and causes infection, pain and the loss of teeth. Choices for managing a carious lesion cover a spectrum of options-from complete surgical excision, where no part of the visible carious tissue is left in the tooth before a restoration is placed, to the opposite extreme, where none of the carious tissue is removed and noninvasive methods are used to prevent progression of the lesion. Thus, this study compared efficacy of no caries removal and sealing the entire lesion verses partial selective caries removal to soft and to firm dentin in healing and/or preventing progression of moderate to deep occlusal dentinal caries in previously unrestored teeth by clinical and radiographic analysis in 4-7 year old children.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age group of 4 - 7 years
* Previously untreated first and second mandibular deciduous molars with moderate to deep occlusal caries i.e. caries involving middle 1/3rd to pulpal 1/3rd of dentin
* No root resorption or physiologic resorption not exceeding 2/3rd of the root length
* Children having positive and definitely positive behavior

Exclusion Criteria:

* Children with special health care needs
* Children with dental crowding limiting the child's ability to maintain oral hygiene
* Teeth with clinical and/or radiological signs or symptoms of non- vitality
* Teeth with clinical and radiological signs or symptoms of irreversible pulpitis or dental abscess (Pain, mobility, tenderness to percussion, draining sinus, pulp polyp, furcal or periapical radiolucency, root resorption)
* Mobility of the tooth
* Pathologic root resorption
* Physiologic root resorption exceeding 2/3rd of root length in preoperative x-ray

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
correlation between caries activity and efficacy of three groups | 12 months
  to check for caries activity and efficacy of three groups i.e. no caries removal, partial caries removal upto soft dentin and partial caries removal upto firm dentin

CONTACTS AND LOCATIONS:
Overall Officials: Sneha D Suwarnkar, MDS, Principal Investigator — Saraswati Dhanwantari Dental College and Hospital, Parbhani
Locations (1):
- Dr Sneha D Suwarnkar, Parbhani, Maharashtra, India